CLINICAL TRIAL: NCT02610192
Title: A Prospective Study of a Single Intra-Articular Injection of Autologous Protein Solution in Females With Primary Patellofemoral Osteoarthritis
Brief Title: nSTRIDE APS in Females With Primary Patellofemoral Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBIO.CR.APSPFO.001.15; APSS-55-00 (Other: Zimmer Biomet)
Record Dates: First submitted 2015-11-10; First posted 2015-11-20 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Patellofemoral Osteoarthritis
Keywords: Autologous Protein Solution; Patellofemoral Osteoarthritis; Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: nSTRIDE Autologous Protein Solution (APS) Kit — Intra-articular injection of APS

SUMMARY:
The purpose of this study is to evaluate clinical outcomes following a single injection of nSTRIDE Autologous Protein Solution in females with isolated patellofemoral osteoarthritis. A secondary objective of this study is to document the duration of treatment effect following nSTRIDE injection.

DETAILED DESCRIPTION:
Clinical trials have, in general, formally demonstrated the effectiveness and safety of various autologous therapies for the treatment of knee OA. Differences in the processing of autologous therapies can yield substantial differences in the resulting output. Thus, making generalizations regarding the effectiveness across these autologous therapies is more complicated. Each autologous therapy requires independent efficacy evaluation. nSTRIDE APS has been shown to decrease pain, increase function and have a favorable safety profile in a pilot trial. Further, demonstration of the treatment effects in patellofemoral osteoarthritis, an important subset of knee osteoarthritis is lacking. This study will evaluate a population of female patients with patellofemoral osteoarthritis in which treatment with other modalities provides limited/short lived relief with the hope that APS treatment will provide and extend relief to these patients. The study will document the treatment effects and timeline of treatment effects for nSTRIDE APS following a single injection (per symptomatic knee).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be female
* Isolated patellofemoral osteoarthritis (PFOA) in one or both knees as diagnosed by the treating physician
* Objective evidence of PFOA on one or both of a radiograph or MRI taken within 3 months of treatment
* From 40-65 years of age, inclusive at time of injection
* Symptoms return such that there is a need for further treatment within 3 months of a corticosteroid or hyaluronic acid injection
* Willing and able to comply with the study procedures
* Sign informed consent form

Exclusion Criteria:

* Any systematic inflammatory condition (e.g. rheumatoid arthritis)
* Active malignancy at time of injection
* Pregnant at time of injection
* Lactating at time of injection
* Knee joint infections or skin diseases or infections in the area of the injection site
* Leukemia, metastatic malignant cells, or who are receiving chemotherapeutic treatment
* Participation in another device, biologic or drug study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verdonk, MD, Principal Investigator — AZ Monica, Deurne
Locations (1):
- AZ Monica, Deurne, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted at a single center in Deurne (Belgium).
Groups:
- nSTRIDE APS: Intra-articular Injection of Autologous Protein Solution (APS)
Period: Overall Study
Arm/Group | nSTRIDE APS
Started | 50 (52 subjects had signed consent form, but 50 subjects have been treated. 2 subjects became SF.)
Completed | 41
Not Completed | 9
Not completed — Received other treatment | 8
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: A total of 52 subjects were enrolled of which 50 subjects were initially treated
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 50.4 (6.5)
Sex/Gender, Customized [Number; unit: participants]
  Gender (female) | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 50

OUTCOME MEASURES:

1. Primary Outcome: Pain Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Subscale Pain at 1, 3, 6 and 12 Months
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's opinion about their knee and associated problems. The original KOOS consists of 5 subscales: Pain (9 questions), Symptoms (7 questions), Function in daily living (ADL) (17 questions), Function in sport and recreation (Sport/Rec) (5 questions) and knee related Quality of Life (QoL) (4 questions). On this scale, 100% indicates no problems and 0% indicates extreme problems.
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 40.3 (18.7)
  1-Month: number analyzed (Participants) | 48
  1-Month | 53.5 (19.8)
  3-Months: number analyzed (Participants) | 45
  3-Months | 52.5 (24.1)
  6-Months: number analyzed (Participants) | 46
  6-Months | 54.9 (22.6)
  12-Months: number analyzed (Participants) | 41
  12-Months | 57.3 (24.8)

2. Secondary Outcome: Symptoms Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Subscale Symptoms at 1, 3, 6 and 12 Months
Description: as for outcome 1
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 46.9 (18.4)
  1-Months: number analyzed (Participants) | 48
  1-Months | 59.2 (19.2)
  3-Months: number analyzed (Participants) | 45
  3-Months | 61.4 (21.6)
  6-Months: number analyzed (Participants) | 46
  6-Months | 61.5 (18.8)
  12-Months: number analyzed (Participants) | 41
  12-Months | 62.5 (22.1)

3. Secondary Outcome: Function in Daily Living (ADL) Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Subscale ADL at 1, 3, 6 and 12 Months
Description: as for outcome 1
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 45.9 (21.1)
  1-Months: number analyzed (Participants) | 48
  1-Months | 58.8 (21.9)
  3-Months: number analyzed (Participants) | 45
  3-Months | 57.9 (26.8)
  6-Months: number analyzed (Participants) | 46
  6-Months | 59.7 (22.8)
  12-Months: number analyzed (Participants) | 41
  12-Months | 62.0 (24.2)

4. Secondary Outcome: Function in Sport and Recreation (Sport/Rec) Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Subscale Sport/Rec at 1, 3, 6 and 12 Months
Description: as for outcome 1
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 11.2 (13.6)
  1-Months: number analyzed (Participants) | 48
  1-Months | 23.0 (20.1)
  3-Months: number analyzed (Participants) | 45
  3-Months | 20.8 (20.2)
  6-Months: number analyzed (Participants) | 46
  6-Months | 22.4 (23.7)
  12-Months: number analyzed (Participants) | 41
  12-Months | 22.9 (24.3)

5. Secondary Outcome: Quality of Life (QoL) Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire Subscale QoL at 1, 3, 6 and 12 Months
Description: as for outcome 1
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 29.7 (10.7)
  1-Months: number analyzed (Participants) | 48
  1-Months | 37.5 (12.1)
  3-Months: number analyzed (Participants) | 45
  3-Months | 37.0 (11.8)
  6-Months: number analyzed (Participants) | 46
  6-Months | 36.3 (13.6)
  12-Months: number analyzed (Participants) | 41
  12-Months | 38.2 (13.5)

6. Secondary Outcome: Pain Measured With Numeric Rating Scales (NRS) Questionnaire Subscale Pain at 1, 3, 6 and 12 Months
Description: The NRS is a validated measure of pain, stiffness and function. The NRS is an 11 point Likert type scale anchored by 0 "no pain" and 10 "worst possible pain". Subjects rate their average pain over the last 24 hours. Likewise subjects rate their stiffness and function on an 11 point Likert type scale
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 6.7 (2.2)
  1-Months: number analyzed (Participants) | 48
  1-Months | 4.9 (2.5)
  3-Months: number analyzed (Participants) | 45
  3-Months | 5.0 (2.9)
  6-Months: number analyzed (Participants) | 46
  6-Months | 4.7 (2.8)
  12-Months: number analyzed (Participants) | 41
  12-Months | 4.5 (2.9)

7. Secondary Outcome: Stifness Measured With Numeric Rating Scales (NRS) Questionnaire Subscale Stiffness at 1, 3, 6 and 12 Months
Description: as for outcome 6
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 6.0 (2.6)
  1-Months: number analyzed (Participants) | 48
  1-Months | 4.3 (2.8)
  3-Months: number analyzed (Participants) | 45
  3-Months | 4.5 (3.1)
  6-Months: number analyzed (Participants) | 46
  6-Months | 4.1 (2.8)
  12-Months: number analyzed (Participants) | 41
  12-Months | 4.0 (3.1)

8. Secondary Outcome: Function Measured With Numeric Rating Scales (NRS) Questionnaire Subscale Function at 1, 3, 6 and 12 Months
Description: as for outcome 6
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 6.6 (2.1)
  1-Months: number analyzed (Participants) | 48
  1-Months | 4.9 (2.4)
  3-Months: number analyzed (Participants) | 45
  3-Months | 4.7 (2.7)
  6-Months: number analyzed (Participants) | 46
  6-Months | 4.7 (2.7)
  12-Months: number analyzed (Participants) | 41
  12-Months | 4.4 (2.9)

9. Secondary Outcome: Patellofemoral Pain and Function Measured With Kujala Anterior Knee Pain Assessment Questionnaire (KAKPAQ) Questionnaire at 1, 3, 6 and 12 Months
Description: The KAKPAQ is a 13-item screening instrument designed to assess patellofemoral pain and instability in adolescents and young adults, with a variable ordinal response format (3-5 choices). The questions included knee functional ability; limping, weight bearing, walking, stairs, squatting, running, jumping, prolonged sitting, pain swelling, painful patellar movement, muscle atrophy and flexion deficiency. Each answer had different scores. To calculate the total score, all items were summarized. The score '0' represented the greatest limitation of knee function, whereas the score '100' indicated the ability to perform most knee functions
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 48.4 (13.0)
  1-Months: number analyzed (Participants) | 48
  1-Months | 55.4 (16.3)
  3-Months: number analyzed (Participants) | 45
  3-Months | 54.8 (17.0)
  6-Months: number analyzed (Participants) | 46
  6-Months | 57.0 (17.0)
  12-Months: number analyzed (Participants) | 41
  12-Months | 56.3 (18.1)

10. Secondary Outcome: Activity Measured With UCLA Activity Score Questionnaire at 1, 3, 6 and 12 Months
Description: The UCLA Activity Score is a validated measure of subject activity. Subjects rate their current activity level from on a simple scale ranging from 1 to 10. The subject indicated her or his most appropriate activity level, with 1 defined as "no physical activity, dependent on others" and 10 defined as "regular participation in impact sports
Time Frame: Baseline, 1, 3, 6 and 12 Months
Population: Analyses were performed on available data, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS
Number analyzed (Participants) | 50
score on a scale
  Baseline | 5.0 (1.9)
  1-Months: number analyzed (Participants) | 48
  1-Months | 5.3 (1.7)
  3-Months: number analyzed (Participants) | 45
  3-Months | 5.5 (2.0)
  6-Months: number analyzed (Participants) | 46
  6-Months | 5.2 (1.8)
  12-Months: number analyzed (Participants) | 41
  12-Months | 5.6 (1.9)

ADVERSE EVENTS:
Time Frame: month 1, month 3, month 6 and month 12
Description: Safety analyses was performed on any knee related AEs, procedure and device related AEs only through 12-Month time point. PLEASE NOTE THAT only knee, procedure, and device related Adverse Events were pre-specified to be collected per protocol. All other AEs were not to be collected within this protocol
Arm/Group | nSTRIDE APS
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nSTRIDE APS (N=50)
Knee Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nSTRIDE APS (N=50)
Excessive Injection Site Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Increased Knee Pain (Musculoskeletal and connective tissue disorders) | 30 (41)
Knee Effusion (Musculoskeletal and connective tissue disorders) | 15 (16)
pain in calf (Musculoskeletal and connective tissue disorders) | 1 (1)
Sprain muscle leg (Musculoskeletal and connective tissue disorders) | 1 (1)
burning feeling lower limb-foot (Musculoskeletal and connective tissue disorders) | 1 (1)
kahler disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — releapse
Stifness (Musculoskeletal and connective tissue disorders) | 6 (8)
fall on knee causing pain (Musculoskeletal and connective tissue disorders) | 3 (3)
inflammation pes anserinus (Musculoskeletal and connective tissue disorders) | 1 (1)
knee twist causing medial bone edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee overload (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain meniscus (Musculoskeletal and connective tissue disorders) | 1 (1)
pain on the medial side due medial root tear (Musculoskeletal and connective tissue disorders) | 1 (1)
worsening OA symptoms (Musculoskeletal and connective tissue disorders) | 1 (1)
wrong movement causing knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT02610192/Prot_SAP_000.pdf